CLINICAL TRIAL: NCT05605275
Title: CRP and PCT as Predictors of Bloodstream Infections in Surgical Patients With Isolation of G+ and G- Bacteria in 3 Year Period
Brief Title: CRP and PCT as Predictors of Sepsis Cause
Status: Completed | Type: Observational
Sponsor: Osijek University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PCT retrospective
Record Dates: First submitted 2022-10-30; First posted 2022-11-04 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2022-10

CONDITIONS: Sepsis; Gram-Positive Bacteremia; Gram-negative Bacteremia
MeSH Terms: conditions — Sepsis | interventions — Leukocyte Count; Platelet Count

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The values of PCT, CRP, white blood cells and platelets will be recorded retrospectively for all patients included in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gram negative: Patients who had at least one blood culture with a gram- isolate during hospitalisation in the surgical ICU
  Interventions: Diagnostic Test: PCT levels; Diagnostic Test: CRP levels; Diagnostic Test: White blood cell count; Diagnostic Test: Platelet count
- Gram positive: Patients who had at least one blood culture with a gram+ isolate during hospitalisation in the surgical ICU
  Interventions: Diagnostic Test: PCT levels; Diagnostic Test: CRP levels; Diagnostic Test: White blood cell count; Diagnostic Test: Platelet count

INTERVENTIONS:
Diagnostic Test: PCT levels — All patients will have their serum PCT level recorded on the day of the positive blood culture and in the next three days.
Diagnostic Test: CRP levels — All patients will have their serum CRP level recorded on the day of the positive blood culture and in the next three days.
Diagnostic Test: White blood cell count — All patients will have their white blood cell (WBC) count recorded on the day of the positive blood culture and in the next three days.
Diagnostic Test: Platelet count — All patients will have their platelets count recorded on the day of the positive blood culture and in the next three days.

SUMMARY:
The aim of this retrospective study is to determine the predictive role of serum level of procalcitonin (PCT) and c-reactive protein (CRP) in determining the causative agent of sepsis in surgical intensive care unit (ICU) patients. The main question it aims to answer is: what serum level of PCT and CRP is predictive of gram+ and gram- sepsis in patients with positive blood cultures in the surgical ICU. The study will be retrospective and will include all patients with positive blood cultures who were hospitalized in the surgical ICU of University Hospital Osijek in the period from January 2019 to May 2022.

DETAILED DESCRIPTION:
PCT is a good biochemical marker of severe bacterial infection. Numerous studies have confirmed its role in the diagnosis of sepsis, especially sepsis with positive blood cultures. This retrospective study will include septic patients who were hospitalised in the surgical ICU between January 2019 and May 2022, and who had at least one positive blood culture. The values of PCT, CRP, white blood cells count and platelets count, as well as the overall outcome of the treatment, will be recorded for the patients included in the research. The aim of the research is to examine the differences in the level of PCT, CRP, white blood cells count and platelets count between patients with gram+ and gram- blood cultures. Also, the predictive value of PCT and CRP in differentiating gram+ from gram- hem will be examined.

ELIGIBILITY:
Inclusion Criteria:

* hospitalisation in surgical ICU
* diagnosis of sepsis
* gram+ blood culture isolate
* gram- blood culture isolate

Exclusion Criteria:

* younger of 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years who were hospitalized in the surgical ICU between January 2019 and May 2022 and who had at least one positive blood culture during treatment will be included in the research.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Predictive level of PCT | 4 days
  Predictive serum level of PCT in differentiating gram+ from gram- blood culture
Predictive level of CRP | 4 days
  Predictive serum level of CRP in differentiating gram+ from gram- blood culture

SECONDARY OUTCOMES:
White blood cells count | 4 days
  Test for differences in WBC count between patients with gram+ and gram- blood cultures
Platelets count | 4 days
  Test for differences in platelets count between patients with gram+ and gram- blood cultures
PCT levels and outcome | 4 days
  To examine differences in serum PCT levels between patients who survived and those who died
CRP levels and outcome | 4 days
  To examine differences in serum CRP levels between patients who survived and those who died

CONTACTS AND LOCATIONS:
Overall Officials: Nenad Neskovic, PhD, Study Chair — Principal Investigator
Locations (1):
- University Hospital Osijek, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morgenthaler NG, Struck J, Fischer-Schulz C, Seidel-Mueller E, Beier W, Bergmann A. Detection of procalcitonin (PCT) in healthy controls and patients with local infection by a sensitive ILMA. Clin Lab. 2002;48(5-6):263-70. PMID 12071576
- [Background] Assicot M, Gendrel D, Carsin H, Raymond J, Guilbaud J, Bohuon C. High serum procalcitonin concentrations in patients with sepsis and infection. Lancet. 1993 Feb 27;341(8844):515-8. doi: 10.1016/0140-6736(93)90277-n. PMID 8094770
- [Background] Sinha M, Desai S, Mantri S, Kulkarni A. Procalcitonin as an adjunctive biomarker in sepsis. Indian J Anaesth. 2011 May;55(3):266-70. doi: 10.4103/0019-5049.82676. PMID 21808399
- [Background] Hoeboer SH, van der Geest PJ, Nieboer D, Groeneveld AB. The diagnostic accuracy of procalcitonin for bacteraemia: a systematic review and meta-analysis. Clin Microbiol Infect. 2015 May;21(5):474-81. doi: 10.1016/j.cmi.2014.12.026. Epub 2015 Jan 14. PMID 25726038
- [Background] Gupta S, Jaswani P, Sharma RK, Agrawal S, Prasad N, Sahu C, Gupta A, Prasad KN. Procalcitonin as a diagnostic biomarker of sepsis: A tertiary care centre experience. J Infect Public Health. 2019 May-Jun;12(3):323-329. doi: 10.1016/j.jiph.2018.11.004. Epub 2018 Nov 26. PMID 30497960
- [Background] Yang L, Lin Y, Wang J, Song J, Wei B, Zhang X, Yang J, Liu B. Comparison of Clinical Characteristics and Outcomes Between Positive and Negative Blood Culture Septic Patients: A Retrospective Cohort Study. Infect Drug Resist. 2021 Oct 12;14:4191-4205. doi: 10.2147/IDR.S334161. eCollection 2021. PMID 34675564